CLINICAL TRIAL: NCT04417166
Title: Pembrolizumab and Radiotherapy for Previously Untreated Patients With Limited Stage NK/T Cell Lymphoma Who Are Not Eligible to Chemotherapy
Brief Title: Pembrolizumab and Radiotherapy for Patients With NK/T Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: International Extranodal Lymphoma Study Group (IELSG) (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IELSG50
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Lymphoma, Extranodal NK-T-Cell
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and Radiotherapy (Experimental): Induction Phase:
  Standard Involved Field Radiation Therapy (IFRT) and pembrolizumab. Pembrolizumab 200 mg IV will be given over 30 minutes on day 1 of each 21 day cycle for a total of 6 cycles. IFRT will start at first cycle of Pembrolizumab and will be delivered concurrently.
  Patients with complete remission (CR), partial response (PR) and stable disease (SD) after Induction Phase will continue with pembrolizumab maintenance.
  Maintenance Phase:
  Pembrolizumab 200 mg IV will be given over 30 minutes on day 1 of each 21 day cycle up to 34 cycles or until disease progression or unaccepted toxicity
  Interventions: Drug: Pembrolizumab; Radiation: Involved Field Radiation Therapy

INTERVENTIONS:
Drug: Pembrolizumab — 50 mg powder for concentrate for solution for infusion
  Other Names: Keytruda
Radiation: Involved Field Radiation Therapy — 50-54 Gy Involved Field Radiation Therapy (IFRT) as proposed by the International Lymphoma Radiation Oncology Group (ILROG) guidelines. 50 Gy is recommended in patients without primary tumor invasiveness (invasion to adjacent tissue and/or organs), 54 Gy in locally advanced cases (invasion to adjacent tissue and/or organs) or with other risk factors (age > 60 years, stage II, elevated serum LDH levels).
  Intensity modulated radiation therapy (IMRT) and volumetric modulated arc therapy (VMAT) are recommended but not mandatory; 3-dimensional conformal RT (3D-CRT) is allowed.

SUMMARY:
Aim of the trial is to evaluate the activity and tolerability of the anti PD1 agent Pembrolizumab in combination with RadioTherapy for the initial treatment of previously untreated patients with limited stage NK/T cell lymphoma who are not eligible to chemotherapy.

It is planned to enroll 30 patients in chinese sites.

All eligible patients will be treated with standard radiotherapy and concurrent pembrolizumab administered intravenously every 3 weeks. After 6 cycles of pembrolizumab patients with complete remission, partial response and stable disease will continue with pembrolizumab maintenance up to 2 years.

Patients will be followed up to 4 years from treatment start.

DETAILED DESCRIPTION:
This is an interventional, phase II, open label, single arm, multicentric clinical trial to be conducted in China.

The primary objective is to test the efficacy of concurrent RT-Pembrolizumab in patients with limited stage NK/T cell lymphoma and who are not eligible to receive chemotherapy.

The secondary objectives are to further explore the efficacy and safety of a the combination of RT and Pembrolizumab as initial treatment of the patients population.

All eligible patients will be treated with standard IFRT and concurrent pembrolizumab administered intravenously, over 30 minutes starting on day 1 of RT (C1D1, at the dose of 200 mg, every 3 weeks). After 6 cycles of pembrolizumab patients will undergo restaging imaging. Patients with complete remission (CR), partial response (PR) and stable disease (SD) will continue with pembrolizumab maintenance up to 2 years that will be administered intravenously, at the dose of 200 mg, over 30 minutes on day 1 every 3 weeks up to 34 cycles.

The follow-up period will last up to 4 years from treatment start.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histological diagnosis of NK/T Cell Lymphoma
* No previous anti-lymphoma treatment
* Age ≥ 18 years
* Ann Arbor stage I-II
* At least one measurable/evaluable site after diagnostic biopsy before treatment start
* At least one of the following high-risk features: age > 60 years, elevated LDH, stage II, primary tumor invasion
* Patient ineligible to receive full dose standard chemotherapy
* ECOG performance status of 0-1
* Signed Informed consent
* Ability to comply with the protocol
* Adequate hematological and organ function;
* Tumor tissue (fresh preferred, archival tissue is also acceptable)
* For women of childbearing potential a negative pregnancy test on day 1 of cycle 1 and agree to adopt an adequate measure to avoid pregnancy during study treatment and for at least one year from end of treatment
* For men agreement to remain abstinent or to use barrier contraception

Exclusion Criteria:

* Advanced stage disease (AA stage III-IV)
* Extranasal type NKTCL
* History of autoimmune disease
* History of other(s) infiltrating cancer(s) in the previous 3 years that were not treated with curative intent or who are still receiving anticancer therapy (including hormone therapy for breast or prostate cancer).
* History of (non-infectious) pneumonitis that required steroids; evidence of interstitial lung disease or active, non-infectious pneumonitis
* Active infection requiring systemic therapy
* Significant cardiovascular disease, myocardial infarction in the previous 3 months, unstable arrhythmias, or unstable angina.
* Prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* HBsAg, HCV or HIV positivity. Positive serology is admitted for HBV and HCV but DNA/RNA test must be negative
* Administration of a live attenuated vaccine within 4 weeks before cyle 1 day 1. Patients must not receive live, attenuate vaccines, including influenza vaccines at any time during study.
* Treatment with systemic immunosuppressive medications, including prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide and anti tumor necrosis factor (anti-TNF) agents within 2 weeks prior to cycle 1 day 1; inhaled corticosteroids are allowed.
* Evidence of suspect of CNS disease
* Clinically significant hypersensitivity (e.g., anaphylactic or anaphylactoid reactions to the compound Pembrolizumab itself or to the excipients in its formulation).
* Has had an allogenic tissue/solid organ transplant
* Known history of active TB (Bacillus Tuberculosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) rate at 2 years - The proportion of patients without disease progression after 2 years from treatment start | 2 years from treatment start
  Response will be assessed using international criteria for response assessment in lymphomas (Cheson 2014) and their update for patients receiving checkpoint inhibitors (Cheson 2016 Lyric)

SECONDARY OUTCOMES:
Complete remission rate (CRR) - Proportion of patients with complete responses | After 4 months from treatment start (End of Induction phase), Maintenance Phase:every 4 months during the first year and then every 6 months until end of treatment. Follow up: every 4 months during first year, then every 6 months during second year
  CRR defined according to Cheson 2014 criteria
2-year Event-free survival - Proportion of patient without disease related events after 2 years from treatment start | 2 years from treatment start
Treatment related mortality - Number of treatment related deaths | From informed consent signature to 90 days after the last study treatment administration
2-year Overall survival - Proportion of patients alive after 2 years from treatment start | 2 years from treatment start
Rate of adverse events - Analysis of incidence, severity and relationship of adverse events | From Informed Consent signature to 30 days for AEs or 90 for SAEs after end of treatment
  Adverse Events severity will be classified according to the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) V. 5.0
Overall Response Rate (ORR) - calculated as the sum of the complete and partial remission rates | After 4 months from treatment start (End of Induction phase) Maintenance Phase: every 4 months during the first year and then every 6 months until end of treatment. Follow up: every 4 months during first year, then every 6 months during second year
  ORR defined according to Cheson 2014 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Luminari, MD, Study Chair — Ematologia, AUSL IRCCS Reggio Emilia; Weili Zhao, MD, Study Chair — Shanghai Rui Jin Hospital,Shanghai Jiao Tong University - School of Medicine
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Shanghai Rui-Jin Hospital, Shanghai